CLINICAL TRIAL: NCT07183904
Title: Analgesic Efficacy of Combined Hematoma and Peripheral Nerve Block Versus Isolated Hematoma Block in the Reduction ff Distal Radius Fractures: A Prospective, Randomized, Multicenter Clinical Trial
Brief Title: Nerve and Hematoma Blocks for Pain Relief During Distal Radius Fracture Reduction
Acronym: BRAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario 12 de Octubre (Other)
Collaborators: Fundación para la Investigación Biomédica Hospital Universitario 12 de Octubre (Unknown)
Responsible Party: Principal Investigator, Jose Antonio Guerrero Serrano, Dr. (Orthopaedic Surgeon), Hospital Universitario 12 de Octubre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24/272
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Acute Distal Radius Fracture; Displaced Distal Radius Fracture
Keywords: Distal Radius Fracture; Hematoma Block; Median Nerve Block; Pain Management; Closed Reduction
MeSH Terms: conditions — Wrist Fractures; Agnosia

STUDY DESIGN:
Intervention Model Description: * Two-arm design with participants randomized 1:1.
  * One group receives hematoma block alone (control).
  * The other group receives hematoma block combined with median nerve block (intervention).
  * Randomization is stratified by study center (Hospital Universitario 12 de Octubre and Hospital Universitario de Getafe) and balanced for sex, age, fracture side, and prior medication use.
  * Each participant is assigned to only one study arm and followed prospectively.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hematoma Block (Active Comparator): Participants will receive a hematoma block only. Under aseptic conditions, 5-10 mL of 2% mepivacaine will be injected directly into the fracture hematoma using a 25-27 gauge needle. No additional nerve block will be performed. This technique is currently the standard of care in the Emergency Department for closed reduction of displaced distal radius fractures.
  Interventions: Procedure: Hematoma Block
- Hematoma Block + Median Nerve Block (Experimental): Participants will receive both a hematoma block and a median nerve block. Median nerve block will be administered at the wrist using anatomical landmarks: 3-5 mL of 2% mepivacaine injected between palmaris longus and flexor carpi radialis.
  Interventions: Procedure: Hematoma Block; Procedure: Median Nerve Block

INTERVENTIONS:
Procedure: Hematoma Block — Injection of 5-10 mL of 2% mepivacaine directly into the fracture hematoma under aseptic conditions.
Procedure: Median Nerve Block — Injection of 3-5 mL of 2% mepivacaine adjacent to the median nerve at the wrist, using anatomical landmarks.
  Arms: Hematoma Block + Median Nerve Block

SUMMARY:
Distal radius fractures, commonly known as wrist fractures, are among the most frequent injuries seen in emergency departments. These injuries often require a closed reduction, a procedure in which the broken bone is manipulated back into place without surgery. One of the main challenges during this procedure is providing adequate pain control.

Traditionally, many hospitals use a "hematoma block," which means injecting a local anesthetic directly into the site of the fracture. This technique is simple and generally safe, but it does not always provide enough pain relief. Some patients continue to experience significant discomfort, especially in the fingers, during the traction and manipulation required to realign the bone.

Another option is to block the median nerve at the wrist. The median nerve supplies sensation to the thumb, index, and middle fingers. When combined with a hematoma block, this technique may improve digital pain relief during fracture reduction. However, this combined approach has not been well studied in Spain, and there is limited high-quality evidence worldwide.

The purpose of this study is to compare two methods of pain control during closed reduction of displaced distal radius fractures in adults: Hematoma block alone versus Hematoma block combined with median nerve block.

We hypothesize that the combined approach will reduce pain more effectively than the hematoma block alone.

The study is designed as a prospective, multicenter, randomized clinical trial involving 112 adult patients treated at two hospitals in Madrid (Hospital Universitario 12 de Octubre and Hospital Universitario de Getafe). Eligible participants are adults aged 18 to 100 years with an acute distal radius fracture (less than 48 hours old) requiring closed reduction. Patients will be randomly assigned to one of the two treatment groups.

Pain will be assessed using a Visual Analog Scale (VAS) at three key moments: during finger traction, during the reduction itself, and at hospital discharge (90-120 minutes after casting). Other information such as age, sex, fracture side, and prior use of pain or psychiatric medication will also be collected.

By answering whether the addition of a median nerve block improves pain control, this study could help establish a new protocol for managing distal radius fractures. If effective, this approach may lead to greater comfort for patients, higher satisfaction, and better overall outcomes in emergency care.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 100 years.
* Diagnosis of acute displaced distal radius fracture (< 48 hours since injury).
* Indication for closed reduction and immobilization.
* Ability to provide informed consent.

Exclusion Criteria:

* Age under 18 years or open physes on plain radiograph.
* Open or pathological distal radius fractures.
* Local infection at or near the planned injection site.
* Significant neurological disease or cognitive impairment interfering with study participation.
* Presence of osteosynthesis material in the same segment of the affected limb.
* Known allergy or contraindication to local anesthetics used in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Pain Intensity During Closed Reduction | During fracture reduction procedure and at hospital discharge (90-120 minutes post-casting).
  Pain will be measured using a 10-cm Visual Analog Scale (VAS, 0 = no pain, 10 = worst imaginable pain). Scores will be recorded at the wrist and fingers during traction, manipulation, and at discharge.

SECONDARY OUTCOMES:
Demographic and Baseline Characteristics | At enrollment (baseline).
  Age, sex, fracture side (left/right), and prior use of analgesic or psychiatric medication will be collected for subgroup analyses.
Incidence of Adverse Events Related to Anesthetic Techniques | From intervention until hospital discharge (90-120 minutes post-casting).
  Documentation of complications such as infection at injection site, hematoma, intravascular injection, systemic anesthetic toxicity (e.g., seizures, arrhythmia), or neuritis.

OTHER OUTCOMES:
Radiographic Quality of Reduction | Immediately after closed reduction and casting.
  Post-reduction radiographs will be evaluated according to the American Academy of Orthopaedic Surgeons (AAOS) and American Society for Surgery of the Hand (ASSH) criteria for acceptable distal radius reduction.

CONTACTS AND LOCATIONS:
Locations (1):
- 12 de Octubre University Hospital, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) collected during the trial that underlie the primary and secondary outcomes will be shared. This includes pain scores (VAS values), demographic information (age, sex, fracture side, prior medication use), and adverse event data. No information that could directly identify a participant (e.g., names, dates of birth, hospital ID numbers) will be included. Requests should be directed to the Principal Investigator (jaguerrero14@hotmail.com)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD Sharing Start Date:
  Approximately 6 months after publication of the primary study results (end-2026).
  IPD Sharing End Date:
  Data will be available for 5 years after publication (end-2031).
Access Criteria: Who will be able to access the IPD and supporting information:
  Qualified researchers with a methodologically sound proposal will be able to access the data. Access will be considered for investigators affiliated with academic institutions or healthcare organizations who intend to use the data for research aligned with the aims of this study.
  What they will be able to access:
  De-identified individual participant data underlying the primary and secondary outcomes (VAS pain scores, demographics, adverse event data), as well as the study protocol, statistical analysis plan, and data dictionary.
  How they will be able to access it:
  Researchers may request access by contacting the Principal Investigator. Following approval of the proposal by the study investigators, the dataset and supporting documents will be transferred using secure, encrypted methods to protect confidentiality.